CLINICAL TRIAL: NCT01078805
Title: Direct Assessment of Non-Vertebral Fractures in Community Experience (DANCE)
Brief Title: Study of FORTEO Use in Subjects in the Community Setting
Acronym: DANCE
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 8492; B3D-US-GHCQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Results first posted 2012-06-26 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-05

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FORTEO (teriparatide)-treated: FORTEO-treated
  Interventions: Drug: FORTEO

INTERVENTIONS:
Drug: FORTEO — prescribed in accordance with usual clinical practice for up to 24 months
  Other Names: Teriparatide; LY333334

SUMMARY:
The purpose of this study is to evaluate the long-term effectiveness, safety, and tolerability of FORTEO in a larger, more diverse "real world" population than studied in clinical trials

DETAILED DESCRIPTION:
Subjects will be followed through a course of FORTEO therapy for up to 24 months and for an additional 24 months after FORTEO treatment is stopped. Subjects may participate in this study for up to 48 months. All aspects of patient care, including diagnostic and therapeutic interventions, will be chosen and conducted at the discretion of the participating study physician according to their clinical judgment and the local standard of medical care.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are judged by the study physician to be suitable for FORTEO therapy. The FORTEO product labeling specifies those individuals diagnosed with osteoporosis who are considered to be at high risk for fracture

Exclusion Criteria:

* Subjects who have an increased baseline risk for osteosarcoma. These include Paget's disease of bone, pediatric populations and young adult patients with open epiphyses, prior external beam or implant radiation therapy involving the skeleton
* Subjects who have administered FORTEO or PTH therapy for more than two weeks directly before study entry
* Subjects who have completed a course of FORTEO or PTH therapy of at least 18 months duration before study entry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 4167 (Actual)
Dates: Start 2003-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakewood, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FORTEO (Teriparatide)-Treated
Started | 4167
Took at Least 1 Dose of Study Drug | 4085
Modified Intent-To-Treat | 3720 (≥1 dose of study drug (SD) and didn't discontinue SD more than 3 consecutive months during treatment)
Completed | 2117
Not Completed | 2050
Not completed — Clinically significant abnormal lab | 5
Not completed — Death | 134
Not completed — Lost to Follow-up | 676
Not completed — Physician Decision | 169
Not completed — Serious adverse event | 26
Not completed — Sponsor decision | 46
Not completed — Withdrawal by Subject | 739
Not completed — Other | 173
Not completed — Didn't take study drug | 82

BASELINE CHARACTERISTICS:
Arm/Group | FORTEO (Teriparatide)-Treated
Number analyzed (Participants) | 3720
Age Continuous [Mean (Standard Deviation); unit: years] | 67.96 (11.72)
Sex/Gender, Customized [Number; unit: participants]
  Female | 3350
  Male | 369
  Unknown | 1
Race/Ethnicity, Customized [Number; unit: participants]
  African | 57
  Asian | 11
  Caucasian | 3282
  East Asian | 29
  Hispanic | 321
  Other | 18
  Unknown | 2
Region of Enrollment [Number; unit: participants]
  United States | 3720
Physician Criteria for Initiating FORTEO Therapy [Number; unit: participants] — Study investigators were provided a questionnaire that was populated with specific criteria they could choose from when they initiated Forteo therapy for their patients. They could have chosen more than one criteria, thus participants could have been counted multiple times. Participants are those who took at least one dose of study drug and had reasons documented to initiate Forteo therapy. The number of total participants analyzed is 4073.
  participants
    New osteoporotic fracture | 848
    Multiple fracture risk factors - per investigator | 3395
    Inadequate response to previous therapy | 2261
    Participant met Forteo threshold -per investigator | 2215
    Intolerance to previous osteoporosis therapy | 891
    Adequate insurance coverage | 925
    Absence of prior authorization criteria | 193
    Participant request | 247
    Height loss | 697

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Non-Vertebral Fragility Fractures
Description: Non-vertebral fragility fracture is defined as low trauma fracture, such as a fall from standing height. It is binary outcome (Yes/No). Percentage of participants = number of participants with new Non-Vertebral Fragility Fracture/ number of participants at risk * 100.
Time Frame: up to 24 months
Population: Participants who received at least one dose of study drug and had non-missing start/stop date, and did not discontinue study drug more than 3 consecutive months at onetime during treatment phase.
Measure: Number; unit: Percentage of participants
Arm/Group | FORTEO (Teriparatide)-Treated
Number analyzed (Participants) | 3720
Percentage of participants
  0 to 6 months (n=3720) | 1.42
  6 to 12 months (n=2970) | 0.91
  12 to 18 months (n=2570) | 0.70
  18 to 24 months (n=2225) | 0.81
Statistical Analysis 1: Comparison: FORTEO (Teriparatide)-Treated; Test type: Superiority or Other; p = 0.0177, One-sample binomial proportion test — Comparison is between 0 to 6 months fracture incidence rate versus 6 to 12 months fracture incidence rate
Statistical Analysis 2: Comparison: FORTEO (Teriparatide)-Treated; Test type: Superiority or Other; p = 0.0019, One-sample binomial proportion test — Comparison is between 0 to 6 months fracture incidence rate versus 12 to 18 months fracture incidence rate
Statistical Analysis 3: Comparison: FORTEO (Teriparatide)-Treated; Test type: Superiority or Other; p = 0.0143, One-sample binomial proportion test — Comparison is between 0 to 6 months fracture incidence rate versus 18 to 24 months fracture incidence rate

2. Secondary Outcome: Percentage of Participants With Clinical Vertebral Fractures
Description: Clinical vertebral fracture was defined as a fracture that caused pain and/or discomfort, came to medical attention, and was confirmed by the investigator. Vertebral fracture sites included thoracic vertebra number 4 (T4) through lumbar spine vertebra number 4 (L4). Vertebral fracture is binary outcome (Yes/No). Percentage of participants= number of participants with new vertebral fracture/ number of participants at risk * 100.
Time Frame: up to 24 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | FORTEO (Teriparatide)-Treated
Number analyzed (Participants) | 3720
Percentage of participants
  0 to 6 months (n=3720) | 0.67
  6 to 12 months (n=2996) | 0.40
  12 to 18 months (n=2606) | 0.35
  18 to 24 months (n=2266) | 0.35
Statistical Analysis 1: Comparison: FORTEO (Teriparatide)-Treated; Test type: Superiority or Other; p = 0.0689, One-sample binomial proportion test — Comparison is between 0 to 6 months fracture incidence rate versus 6 to 12 months fracture incidence rate
Statistical Analysis 2: Comparison: FORTEO (Teriparatide)-Treated; Test type: Superiority or Other; p = 0.0412, One-sample binomial proportion test — Comparison is between 0 to 6 months fracture incidence rate versus 12 to 18 months fracture incidence rate
Statistical Analysis 3: Comparison: FORTEO (Teriparatide)-Treated; Test type: Superiority or Other; p = 0.0631, One-sample binomial proportion test — Comparison is between 0 to 6 months fracture incidence rate versus 18 to 24 months fracture incidence rate

3. Secondary Outcome: Percentage Change From Baseline in Back Pain Score by Visual Analog Scale (VAS) at 24 Month Endpoint
Description: Visual analog pain scale is a measurement instrument to measure the level of pain. Scores range from 0 to 100. Higher score indicates greater pain. Mean percentage change is (Pain score at baseline visit - Pain score at Month 24)/Pain score at baseline visit*100%.
Time Frame: Baseline, Month 24
Population: Participants with at least a VAS score of 40 at baseline and at least one post-baseline measurement.
Measure: Mean (Standard Error); unit: percentage change of pain score
Arm/Group | FORTEO (Teriparatide)-Treated
Number analyzed (Participants) | 289
percentage change of pain score | -36.2 (2.8)
Statistical Analysis 1: Comparison: FORTEO (Teriparatide)-Treated; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

4. Secondary Outcome: Percentage Change From Baseline in Pain Score by Visual Analog Scale (VAS) at 24 Month Endpoint
Description: as for outcome 3
Time Frame: Baseline, Month 24
Population: Participants with at least a VAS score of 40 at baseline and at least one post-baseline measurement.
Measure: Mean (Standard Error); unit: percentage change of pain score
Arm/Group | FORTEO (Teriparatide)-Treated
Number analyzed (Participants) | 375
percentage change of pain score | -24.9 (2.2)
Statistical Analysis 1: Comparison: FORTEO (Teriparatide)-Treated; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

5. Secondary Outcome: Treatment Adherence
Description: Treatment adherence is the duration of time participants were on Forteo therapy during the 24-month treatment phase of the study.
Time Frame: up to 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FORTEO (Teriparatide)-Treated
Number analyzed (Participants) | 3720
days
  0 to 6 months (n=701) | 72.5 (54.5)
  6 to 12 months (n=382) | 272.5 (57.7)
  12 to 18 months (n=338) | 450.7 (59.0)
  18 to 24 months (n=2299) | 743.7 (115.7)

6. Secondary Outcome: Percentage Change From Baseline in Bone Mineral Density (BMD) at Month 24 Endpoint
Description: A BMD test measures the amount of mineral (such as calcium) in a defined area of bone, grams per square centimeter (g/cm²).
Time Frame: Baseline, up to month 24
Population: Participants who received at least one dose of study drug and had non-missing start/stop date, and did not discontinue study drug more than 3 consecutive months at onetime during treatment phase. At least one post-baseline measurement within 24 month, last observation carried forward.
Measure: Mean (Standard Error); unit: percentage (%) change of BMD
Arm/Group | FORTEO (Teriparatide)-Treated
Number analyzed (Participants) | 835
percentage (%) change of BMD
  Femoral Neck | 2.569 (0.944)
  Forearm | 0.626 (1.421)
  Inter-Trochanter | 1.532 (0.413)
  Lumbar spine vertebrae numbered 1 through 4(L1-L4) | 6.419 (0.334)
  Total Hip | 3.766 (1.721)
  Trochanter | 2.604 (1.186)
  Wards Triangle | 3.394 (0.761)

7. Secondary Outcome: Percentage Change From Baseline in Bone Mineral Content (BMC) at Month 24 Endpoint
Description: BMC is an estimate of the amount of mineral (such as calcium) in the bone.
Time Frame: Baseline, up to month 24
Population: as for outcome 6
Measure: Mean (Standard Error); unit: percentage (%) change of grams (g)
Arm/Group | FORTEO (Teriparatide)-Treated
Number analyzed (Participants) | 590
percentage (%) change of grams (g)
  Femoral Neck | 4.187 (1.707)
  Forearm | 7.243 (7.995)
  Inter-Trochanter | 5.716 (2.684)
  L1-L4 | 20.774 (11.226)
  Total Hip | 8.303 (6.866)
  Trochanter | 4.968 (2.899)
  Wards Triangle | 50.996 (30.540)

8. Secondary Outcome: Percentage Change From Baseline in Bone Area at Month 24 Endpoint
Description: Bone area is a defined region of interest of bone.
Time Frame: Baseline, up to month 24
Population: as for outcome 6
Measure: Mean (Standard Error); unit: percent change of centimeter square
Arm/Group | FORTEO (Teriparatide)-Treated
Number analyzed (Participants) | 591
percent change of centimeter square
  Femoral Neck | 2.231 (1.336)
  Forearm | 4.680 (4.705)
  Inter-Trochanter | 1.828 (0.661)
  L1-L4 | 3.907 (1.242)
  Total Hip | 2.648 (1.453)
  Trochanter | 3.395 (2.375)
  Wards Triangle | 1.826 (1.171)

9. Secondary Outcome: Physician Criteria for Initiating FORTEO Therapy
Description: Study investigators were provided a questionnaire that was populated with specific criteria they could choose from when they initiated Forteo therapy for their patients. They could have chosen more than one criteria, thus participants could have been counted multiple times. As this was actually a baseline characteristic rather than an outcome measure, data are presented in the baseline characteristic table rather than here.
Time Frame: Baseline
Population: Participants are those who took at least one dose of study drug and had reasons documented to initiate Forteo therapy. This is a baseline characteristic; therefore data are presented in the section of Baseline Characteristics.
Measure: Number; unit: participants
Arm/Group | FORTEO (Teriparatide)-Treated
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Per Protocol, this study only required the collection of serious adverse events (SAEs). SAEs were collected during the entire treatment phase plus 30 days after cessation of Forteo treatment, and if the SAE was deemed related to Forteo treatment during the cessation phase.
Arm/Group | FORTEO (Teriparatide)-Treated
Serious Adverse Events (participants affected / at risk) | 432/4085
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FORTEO (Teriparatide)-Treated (N=4085)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Spleen disorder (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2)
Arteriospasm coronary (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 11 (11)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 3 (3)
Cardiac disorder (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 10 (10)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 4 (4)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Coronary artery perforation (Cardiac disorders) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 18 (18)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Right ventricular failure (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 4 (4)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 2 (2)
Goitre (Endocrine disorders) | 1 (1)
Amaurosis fugax (Eye disorders) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Acute abdomen (Gastrointestinal disorders) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1)
Femoral hernia (Gastrointestinal disorders) | 1 (1)
Femoral hernia, obstructive (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 2 (2)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Intestinal infarction (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 5 (5)
Intestinal strangulation (Gastrointestinal disorders) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 14 (14)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Asthenia (General disorders) | 2 (2)
Chest pain (General disorders) | 10 (10)
Chills (General disorders) | 1 (1)
Death (General disorders) | 15 (15)
Device occlusion (General disorders) | 1 (1)
Hernia (General disorders) | 1 (1)
Impaired healing (General disorders) | 1 (1)
Medical device complication (General disorders) | 3 (3)
Multi-organ failure (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Sudden death (General disorders) | 2 (2)
Biliary cirrhosis primary (Hepatobiliary disorders) | 1 (1)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 4 (4)
Cholecystitis acute (Hepatobiliary disorders) | 5 (5)
Cholelithiasis (Hepatobiliary disorders) | 4 (4)
Chronic hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatic congestion (Hepatobiliary disorders) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1)
Acquired immunodeficiency syndrome (Infections and infestations) | 1 (1)
Anogenital warts (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2)
Appendicitis perforated (Infections and infestations) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 6 (6)
Bronchitis bacterial (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 2 (2)
Catheter site infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 7 (7)
Clostridial infection (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (2)
Device related infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 4 (4)
Endocarditis (Infections and infestations) | 1 (1)
Gastric infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 4 (4)
Influenza (Infections and infestations) | 2 (2)
Kidney infection (Infections and infestations) | 2 (2)
Labyrinthitis (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Lung infection pseudomonal (Infections and infestations) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 2 (2)
Peritonitis bacterial (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 37 (37)
Pneumonia haemophilus (Infections and infestations) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 4 (4)
Septic shock (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1)
Small intestine gangrene (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 3 (3)
Streptococcal infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 13 (13)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 3 (3)
Viral infection (Infections and infestations) | 2 (2)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 4 (4)
Compression fracture (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 38 (38)
Femur fracture (Injury, poisoning and procedural complications) | 9 (9)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 22 (22)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 2 (2)
Pelvic fracture (Injury, poisoning and procedural complications) | 4 (4)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Pseudomeningocele (Injury, poisoning and procedural complications) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2)
Sternal fracture (Injury, poisoning and procedural complications) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 4 (4)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 5 (5)
Tibia fracture (Injury, poisoning and procedural complications) | 4 (4)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 5 (5)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2)
Blood pressure decreased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Bone scan abnormal (Investigations) | 1 (1)
Heart rate increased (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Light chain analysis increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 10 (10)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2)
Haemochromatosis (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 (11)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 (2)
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 2 (2)
Brain oedema (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 12 (12)
Convulsion (Nervous system disorders) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Dysarthria (Nervous system disorders) | 1 (1)
Encephalitis (Nervous system disorders) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (3)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1)
Multiple sclerosis relapse (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Radicular pain (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 7 (7)
Transient ischaemic attack (Nervous system disorders) | 5 (5)
Agitation (Psychiatric disorders) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Hallucination (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Pyuria (Renal and urinary disorders) | 1 (1)
Renal amyloidosis (Renal and urinary disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 6 (6)
Renal failure acute (Renal and urinary disorders) | 5 (5)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 2 (2)
Adenomyosis (Reproductive system and breast disorders) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1)
Pelvic prolapse (Reproductive system and breast disorders) | 2 (2)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1)
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 16 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Pulmonary eosinophilia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Colectomy (Surgical and medical procedures) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Medical device removal (Surgical and medical procedures) | 1 (1)
Shoulder arthroplasty (Surgical and medical procedures) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1)
Aortic aneurysm (Vascular disorders) | 4 (4)
Aortic stenosis (Vascular disorders) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 6 (6)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (5)
Hypotension (Vascular disorders) | 2 (2)
Intermittent claudication (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 4 (4)
Superior mesenteric artery syndrome (Vascular disorders) | 1 (1)
Venous insufficiency (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days